CLINICAL TRIAL: NCT03406091
Title: Detection of Poor Mobilizer (PM) in Multiple Myeloma (MM) Patients: Prospective Product Registry
Brief Title: Detection of Poor Mobilizer (PM) in Multiple Myeloma (MM) Patients
Status: Completed | Type: Observational
Sponsor: Fondazione EMN Italy Onlus (Other)
Responsible Party: Sponsor
Other Study IDs: MOZOBL06877
Record Dates: First submitted 2018-01-15; First posted 2018-01-23 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — plerixafor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Poor Mobilizer (PM) in Multiple Myeloma (MM) patients
  Interventions: Drug: Plerixafor

INTERVENTIONS:
Drug: Plerixafor — Plerixafor (AMD3100) is a selective, reversible inhibitor of the receptor chemokine (C-X-C motif) receptor 4 (CXCR4) and prevents binding of its cognate ligand stromal cell derived factor-1α (SDF-1α), also known as chemokine (C-X-C motif) ligand 12 (CXCL12) [3]. CXCR4 is a co-receptor, along with CD4, for the binding of human immunodeficiency virus, type 1 (HIV-1) to its receptor cells.

SUMMARY:
The study is an italian multicentric and will be conducted in 20 centers. The aim of this study is to evaluate poor mobilizer (PM) rate in newly diagnosed MM patients who are mobilized with cyclophosphamide and G-CSF and plerixafor on demand.

Plerixafor is a specific reversible inhibitor of the chemokine receptor CXCR4 and prevents the binding of its ligand stromal cell derived factor SDF-1α also known as CXCL12, thereby releasing hematopoietic stem cells into the circulation.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed transplant eligible MM patients
2. Measurable disease as defined by the presence of M-protein in serum or urine, or abnormal free light chain ratio
3. Eligible and planned for HDT and autologous haematopoietic stem cell transplantation
4. ≥18 years of age
5. Patients or their legally authorized representatives must provide written informed consent
6. Mobilization performed with G-CSF 2-4 g/m2 of cyclophosphamide and Plerixafor On Demand if considered needed based on center policies
7. Patients can be included in interventional clinical trials
8. Karnofsky performance status ≥ 60%
9. Total bilirubin < 1.5 upper limit of normal (ULN)
10. AST/SGOT and ALT/SGPT < 2.5 upper limit of normal (ULN)
11. Serum creatinine < 2 upper limit of normal (ULN)
12. WBC count ≥2.5x109/L
13. ANC count ≥1.5x109/L
14. Platelet count ≥75x109/L
15. Adequate cardiac, renal, and pulmonary function sufficient to undergo apheresis and transplantation, i.e., eligible by institutional standards for autologous stem cell transplant
16. Women are not breast feeding and not pregnant
17. A negative pregnancy test is required for women in child-bearing age; patients must agree to use an adequate method of contraception whilst on study treatment and for 3 months following plerixafor treatment

Exclusion Criteria:

1. Relapse/refractory MM patients
2. Non secretory MM
3. Primary plasmacell leukemia.
4. Age < 18.
5. Prior allogeneic or autologous transplantation.
6. Prior failed mobilization attempt.
7. Inability to tolerate PBPC harvest.
8. Peripheral venous access not possible.
9. Pregnant or nursing women or patients unwilling to have adequate contraception up to 3 months after end of treatment with plerixafor
10. Clinical active infectious hepatitis type A, B, C or HIV
11. Acute infection (febrile, i.e. temperature > 38°C) within 24 hours prior to dosing or antibiotic therapy within 7 days prior to the first dose of GCSF.
12. Left ventricular ejection fraction < 50%.
13. Splenectomised or splenic irradiation.
14. Psychiatric, addictive, or any disorder/disease which compromises ability to give truly informed consent for participation in this study and renders the patient at high risk from treatment complications or impairs the ability to comply with the study treatment and protocol.
15. Treatment with G-CSF or other cytokine within 2 weeks prior to the first dose of G-CSF for mobilization.
16. Patients previously treated with Plerixafor
17. Patients mobilised with chemotherapy other than cyclophosphamide 2 et 4 gr/m2
18. Patients mobilised with growth factors at a dose other than (5-10µg/kg)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 300 eligible patients ≥18 years old diagnosed with MM who are eligible to undergo treatment with an autologous haematopoietic stem cell transplant may be enrolled. Patients must meet all the inclusion criteria listed below within 7 days of first administration of cyclophosphamide in addition to signing an informed consent form.
  A patient will be considered enrolled after he/she has met all eligibility criteria and has started the protocol treatment.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2015-11-26 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Assessment of success rate expressed as % of patients mobilizing ≥2x106 CD34+ cells/kg in maximum 3 apheresis and patient who achieves the optimal target of 4x106 CD34+ cells/kg up to 5 apheresis. | 3 years

SECONDARY OUTCOMES:
% of patients having received plerixafor in the study population | 3 years
Evaluate in patients failing mobilisation how many of them received plerixafor and how many did not | 3 years
Evaluation of speed of mobilization using plerixafor, in terms of increase in number of circulating CD34+ cells from time 0 to 6-11 hours after the first dose of plerixafor. | 3 years
Total number of CD34+ cells collected per apheresis day | 3 years
Confirmation of factors predicting a poor mobilization: patients who experienced grade 3-4 haematological toxicity during induction, used lenalidomide as induction treatment, aged > 60 years old and experienced cytopenia at diagnosis. | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- A.O.U. Città della Salute e della Scienza di Torino, Torino, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mina R, Petrucci MT, Bonello F, Bongarzoni V, Saccardi R, Bertuglia G, Mengarelli A, Spadaro A, Lisi C, Curci P, Lemoli RM, Ballanti S, Floris R, Cupelli L, Tosi P, Olivieri A, Rota-Scalabrini D, Cangialosi C, Nozzoli C, Anaclerico B, Fazio F, Bruno B, Mancuso K, Corradini P, Milone G, Boccadoro M. A prospective, multicenter study on hematopoietic stemcell mobilization with cyclophosphamide plus granulocyte colony-stimulating factor and 'on-demand' plerixafor in multiple myeloma patients treated with novel agents. Haematologica. 2024 May 1;109(5):1525-1534. doi: 10.3324/haematol.2023.284023. PMID 37981892